CLINICAL TRIAL: NCT06920693
Title: A Phase 1, First in Human, Randomised, Double-Blind, Placebo-controlled, Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) Study to Investigate the Safety, Tolerability and Pharmacokinetics of GB-7624 Administered Subcutaneously in Healthy Adult Participants
Brief Title: Study to Investigate the Safety, Tolerability, and Pharmacokinetics of GB-7624 in Healthy Adult Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Generate Biomedicines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB-7624-101
Record Dates: First submitted 2025-03-11; First posted 2025-04-10 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study intervention: GB-7624 (Experimental)
  Interventions: Drug: GB-7624
- Study Intervention: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB-7624 — Study Drug GB-7624
  Arms: Study intervention: GB-7624
Drug: Placebo — Placebo
  Arms: Study Intervention: Placebo

SUMMARY:
This is a randomised, double-blinded, placebo-controlled first in human (FIH) trial to evaluate the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD), and immunogenicity of GB-7624. The trial will have two parts: a SAD component and a MAD component.

Part A (SAD): a total of 24 healthy volunteers are planned to be enrolled across 3 SAD cohorts and will involve the administration of a single subcutaneous (SC) dose of GB-7624 (300 mg, 600 mg, or 1200 mg) or placebo on Day 1 in cohorts A1, A2, and A3.

Part B (MAD): a total of 16 healthy volunteers are planned to be enrolled across 2 MAD cohorts and will involve the administration of multiple SC doses of GB-7624 (300 mg on Day 1 and Day 15 or 600 mg on Day1 and Day 15) or placebo in cohorts B1 and B2.

The decision to escalate between dose levels in the SAD (Part A) and the MAD (Part B) as well as the decision to proceed from Part A to Part B will be based on safety review committee (SRC) review of prior cohorts, blinded available safety, tolerability and PK data.

Study drug will be administered at the study site by trained study site personnel to ensure compliance. The administration of all trial intervention will be recorded in eCRF. Compliance will be assured by direct supervision and witnessing of trial intervention administration.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have given written informed consent before any trial-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.
2. Adults, 18 to 65 years of age (inclusive) at the screening visit.
3. Body mass index (BMI) greater than or equal to 18.0 and less than or equal to 32.0 kg/m2 (inclusive)
4. Medically healthy as determined by medical history, vital signs, physical examination (no CS findings),ECG and clinical laboratory tests at screening and pre-dose on Day -1 or Day 1. This includes the following:

   1. Systolic blood pressure (BP) in the range of 90 to 140 mmHg (inclusive) and diastolic BP in the range of4050 to 90 mmHg (inclusive) after 5 minutes in seated, semi-recumbent, or supine position
   2. Heart rate (HR) in the range of 40 to 100 bpm (inclusive) after 5 minutes rest in seated, semi-recumbent, or supine position
   3. Body temperature, between 35.5°C and 37.5°C (inclusive)
   4. Electrocardiogram (ECG) without CS abnormalities including QT interval corrected for Fredericia (QTcF) <450 msec for male participants and <470 msec for female participants.
   5. In the opinion of the investigator, no significant findings in serum chemistry, haematology, coagulation and urinalysis tests.
5. Female volunteers must:

   1. Be of non-child-bearing potential i.e., surgically sterilised (hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 6 months before the screening visit or postmenopausal (where postmenopausal is defined as no menses for 12 months without an alternative medical cause and a follicle-stimulating hormone (FSH) level consistent with postmenopausal status, per local laboratory guidelines), or
   2. A woman of childbearing potential (WOCBP) must have a negative pregnancy test at Screening (blood test) and before the first trial drug administration (Day -1 urine test). They must agree not to attempt to become pregnant or donate ova and to use protocol-defined methods of contraception from one month prior to screening until at least 360 days after the last dose of study drug.
   3. Women who are currently lactating, breastfeeding, receiving hormone therapy with the intention of having children, planning to donate ova or planning to become pregnant during the trial and within 360days after last dose of trial drug, are excluded from participation.
6. Male participants (including vasectomised males and those with documented azoospermia): must agree to not donate sperm and, if engaging in sexual intercourse with a WOCBP, must agree to use a condom in addition to using use protocol-defined methods of contraception and agree to refrain from donating sperm from screening through at least 360 days after the last dose of trial drug. If engaging in sexual intercourse with a female partner who is not of childbearing potential or a same-sex partner, agree to use a condom from signing the consent form until at least 360 days after the last dose of study drug.
7. Have suitable venous access for blood sampling.
8. Be willing and able to comply with all trial assessments and adhere to the protocol schedule and restrictions

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary (excluding resolved childhood asthma, at the discretion of the PI or delegate), hepatic, renal, haematological, neoplastic, gastrointestinal, endocrine, immunologic, dermatologic, neurological (excluding migraine, at the discretion of the PI or delegate),ocular or psychiatric disease (excluding non-hospitalised depression and anxiety, at the discretion of the PI or delegate), including any acute illness or surgery within the past 3 months determined by the PI (in consultation with the MM/SMR) to be clinically relevant. Participants with a history of malignant disease in the last 5 years (excludes localised, non-melanoma skin cancers treated with curative intent and not on active therapy).
2. Current infection or acute illness or fever within 3 days before trial enrolment (enrolment may be delayed for full recovery if acceptable to the investigator), that requires antibiotic, antifungal or antiviral medications.
3. Diagnosed active helminth infection or travel in last 3 months to areas at high risk of these infections.
4. Positive testing for human immunodeficiency virus (HIV)-1 and 2, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) antibodies at the screening visit.
5. Current smokers or ex-smokers who have given up smoking for less than or equal to 3 months. Social/casual smokers (defined as <5 cigarettes per week) may be included if willing to completely abstain from smoking from screening through the duration of the trial.
6. Positive cotinine testing at Day -1.
7. Presence or history of substance abuse, alcohol abuse or excessive intake of alcohol within 2 years prior to screening (refer to exclusion criterion 9 and 10).
8. Positive coronavirus disease 2019 (COVID-19) test on Day -1.
9. Positive drug or alcohol testing at screening and/or Day -1.
10. Regular consumption of more than 10 standard alcoholic drinks/week and/or more than 4 standard alcoholic drinks on any one day, where 1 standard drink is 10 g of pure alcohol and is equivalent to 285 mL beer [4.9% Alc/Vol], 100 mL wine [12% Alc/Vol], or 30 mL spirit [40% Alc/Vol]).
11. History of any severe allergic reactions (necessitating hospitalisation, oxygen and/or epinephrine use),which in the opinion of the PI (or delegate), would interfere with the volunteer's ability to participate in the study.
12. Use of any prescription within 14 days prior to admission to the study site (Day -1) and/or non-prescription, over-the-counter (OTC) medication (including dietary or herbal supplements) within 7 days or 5 half-lives of the medication (whichever is longer) prior to admission to the study site (Day -1), except use of contraceptives or hormone replacement therapy and the use of paracetamol (up to 2 g per day).Vitamins may be permitted in discussion with the Sponsor.
13. History of risk factors for torsade de pointes (including a family history of long QT syndrome or sudden cardiac death) or a known arrythmia.
14. Liver function test results elevated >1.5-fold above the upper limit of normal (ULN) for bilirubin (total, conjugated and unconjugated), alkaline phosphatase (ALP), aspartate aminotransferase (AST) or alanine aminotransferase (ALT).
15. Estimated creatinine clearance (CrCl) < 60 mL/min using the Cockcroft-Gault formula or serum creatinine >1.5-fold above the ULN.
16. History of sensitivity to any of the trial medications, or its components, or a history of drug reaction or other allergies that, in the opinion of the PI or MM, contradict their participation.

    Note: This includes any previous allergic reaction to biologic agents.
17. Presence or evidence of recent sunburn, scar tissue, tattoos, open sores, or dermatological conditions, that in the opinion of the PI (or delegate) would interfere with the intended SC injection site or evaluation of the participant's response to the study drug and ability to assess for any injection site reactions.
18. Receipt of any live attenuated vaccinations within 30 days prior to admission to the study site (Day -1)and non-live vaccines within 14 days prior to admission to the study site (Day -1).

    Note: Influenza, COVID-19 and pneumococcal vaccines permitted up to 7 days prior to admission to the study site (Day -1).
19. Donation of whole blood within 30 days prior to admission to the study site (Day -1), or loss of whole blood of more than 500 mL within 30 days prior to admission to the study site (Day -1). Receipt of a bloodtransfusion within 1 year of the admission to the study site (Day -1).
20. Donation of plasma within 1 week prior to screening visit.
21. Receipt of any biological drugs such as monoclonal antibodies, immunoglobulin or other bloodproducts within 3 months or 5 half-lives (whichever is longer) of admission to the study site (Day -1).
22. Participation in another investigational clinical trial with the EOS visit for the trial within 30 days prior toadmission to the study site (Day -1) or within 5 half-lives of the previous investigational drug (whichever islonger).
23. Any other condition or prior therapy, which, in the opinion of the PI, would make the participant unsuitable for this trial, including unable to cooperate fully with the requirements of the trial protocol or likely to be non-compliant with any trial requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite Outcome: To assess the safety and tolerability of single doses of GB-7624 administered subcutaneously (SC) in healthy volunteers. | Day -1 to Day 360
  Participant incidence and severity of treatment-emergent adverse events (TEAEs), serious AEs (SAEs),and TEAEs leading to discontinuation of study treatment.
  Clinically significant (CS) changes from baseline in:
  * Clinical laboratory results (haematology, clinical chemistry, coagulation and urinalysis)
  * Vital signs
  * Twelve-lead electrocardiograms (ECGs)
Composite Outcome: To assess the safety and tolerability of multiple doses of GB-7624 administered SC in healthy volunteers | Day -1 to Day 360
  Participant incidence and severity of treatment-emergent AEs (TEAEs), serious AEs (SAEs), and TEAEs leading to discontinuation of study treatment.
  Clinically significant (CS) changes from baseline in:
  * Clinical laboratory results (haematology, clinical chemistry, coagulation and urinalysis)
  * Vital signs
  * Twelve-lead electrocardiograms (ECGs)

SECONDARY OUTCOMES:
To characterise the maximum concentration (Cmax) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The Cmax of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the time to peak drug concentration (Tmax) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The Tmax of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the half-life (t1/2) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The t1/2 of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the the area under the curve to last quantifiable timepoint (AUClast) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUClast of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the volume of distribution (V/F) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The V/F of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the the area under the plasma concentration-time curve (AUC) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUC of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the the area under the plasma concentration-time curve from time zero to infinity (AUCinf) of GB-7624 following single doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUCinf of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the total body clearance from plasma (CL/F) of GB-7624 following singles dose of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The CL/F of GB-7624 following single SC doses in healthy volunteers will be analyzed
To characterise the maximum concentration (Cmax) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The Cmax of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the time to peak drug concentration (Tmax) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The Tmax of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the half-life (t1/2) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The t1/2 of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the the area under the curve to last quantifiable timepoint (AUClast) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUClast of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the volume of distribution (V/F) of GB-7624 following a multiple dose of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The V/F of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the the area under the plasma concentration-time curve (AUC) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUC of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the the area under the plasma concentration-time curve from time zero to infinity (AUCinf) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The AUCinf of GB-7624 following multiple SC doses in healthy volunteers will be analyzed
To characterise the total body clearance from plasma (CL/F) of GB-7624 following multiple doses of GB-7624 administered SC in healthy volunteers | Day 1 to Day 360
  The CL/F of GB-7624 following multiple SC doses in healthy volunteers will be analyzed

CONTACTS AND LOCATIONS:
Locations (1):
- Generate Biomedicines Clinical Site, Herston, Queensland, Australia